CLINICAL TRIAL: NCT06663319
Title: A Phase I Study of JNJ-89402638 for Unresectable Metastatic Colorectal Cancer
Brief Title: A Study of JNJ-89402638 for Metastatic Colorectal Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 89402638GIC1001; 89402638GIC1001 (Other: Janssen Research & Development, LLC); 2024-516526-66-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2024-10-28; First posted 2024-10-29 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Unresectable Metastatic Colorectal Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- JNJ-89402638 (Experimental): Participants with unresectable metastatic colorectal adenocarcinoma (mCRC) will receive JNJ-89402638 in Part 1 (Dose escalation) of the study and the dose levels will be escalated sequentially until the recommended Phase 2 Dose(s) (RP2D) have been identified. Participants in Part 2 (Dose expansion) will receive JNJ-89402638 at the RP2D(s) determined in Part 1.
  Interventions: Drug: JNJ-89402638

INTERVENTIONS:
Drug: JNJ-89402638 — JNJ-89402638 will be administered.

SUMMARY:
The purpose of this study is to determine the putative recommended phase 2 dose(s) (RP2Ds) of JNJ-89402638 and to determine the safety of JNJ-89402638 at the RP2D(s) in participants with metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically or cytologically confirmed diagnosis of colorectal adenocarcinoma (CRC) progressing after 2 or more prior lines of standard therapy in the metastatic/unresectable setting
* Have evaluable or measurable disease per response evaluation criteria in solid tumors (RECIST) version 1.1

  1. Part 1: Must have either measurable or evaluable disease
  2. Part 2: Must have at least 1 measurable lesion
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Have an estimated or measured glomerular filtration rate (GFR) greater than or equal to (>=) 30 milliliter per minute (mL/min) based on modification of diet in renal disease (MDRD) 4-variable formula

Exclusion Criteria:

* Active (new or progressive) brain metastases, leptomeningeal disease, or untreated spinal cord compression
* Toxicity from prior anticancer therapy that has not resolved to Grade less than or equal to (<=)1 (except alopecia, vitiligo, Grade <= 2 peripheral neuropathy, or endocrinopathies that are stable on hormone replacement)
* Has a prior or concurrent second malignancy (other than the disease under study) unless natural history or treatment is unlikely to interfere with any study endpoints of safety or the efficacy of the study treatment
* Received glucocorticoids (doses >10 mg/day prednisone or equivalent) within 7 days prior to the first dose of study drug
* Received or plans to receive any live, attenuated vaccine within 4 weeks before the first dose of study treatment or within 4 weeks after the last dose of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2028-02-25 (Estimated); Study Completion 2028-07-19 (Estimated)

PRIMARY OUTCOMES:
Part 1 and Part 2: Number of Participants with Adverse Events (AEs) by Severity | From Baseline up to approximately 24 months
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Severity of AEs will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. Cytokine release syndrome (CRS) and immune effector cell-associated neurotoxicity syndrome (ICANS) will be graded per American Society for Transplantation and Cellular Therapy (ASTCT) consensus.
Part 1: Number of Participants with Dose-Limiting Toxicity (DLT) | From Baseline up to 28 days
  The DLTs are specific adverse events including high grade hematologic or non-hematologic toxicities.

SECONDARY OUTCOMES:
Part 1 and Part 2: Serum Concentration for JNJ-89402638 | Up to approximately 24 months
  Serum Concentration for JNJ-89402638 will be reported.
Part 1 and Part 2: Maximum Serum Concentration (Cmax) of JNJ-89402638 | Up to approximately 24 months
  Cmax of JNJ-89402638 will be reported.
Part 1 and Part 2: Minimum Serum Concentration (Cmin) of JNJ-89402638 | Up to approximately 24 months
  Cmin of JNJ-89402638 will be reported.
Part 1 and Part 2: Time to Reach Maximum Observed Serum Concentration (Tmax) of JNJ-89402638 | Up to approximately 24 months
  Tmax of JNJ-89402638 will be reported.
Part 1 and Part 2: Area Under the Serum Concentration-time Curve (AUC) of JNJ-89402638 | Up to approximately 24 months
  AUC of JNJ-89402638 will be reported.
Part 1 and Part 2: Number of Participants with Presence of Anti-JNJ-89402638 Antibodies | Up to approximately 24 months
  Participants with anti-JNJ-89402638 antibodies will be reported.
Part 1 and Part 2: Overall Response (OR) | Up to approximately 24 months
  Overall response is best response of complete response (CR) or partial response (PR), assessed according to response evaluation criteria in solid tumors (RECIST) version 1.1.
Part 1 and Part 2: Complete Response (CR) | Up to approximately 24 months
  Complete response is defined as a best response of CR assessed according to RECIST version 1.1.
Part 1 and Part 2: Time to Response (TTR) | Up to approximately 24 months
  TTR is defined for participants who achieved an OR from the time of the first dose of study treatment to the first response of PR or better as assessed according to RECIST version 1.1.
Part 1 and Part 2: Duration of Response (DOR) | Up to approximately 24 months
  DOR is defined for participants who achieved an OR in the time between the date of initial documentation of first response of PR or better to the date of first documented evidence of progressive disease or death due to any cause, whichever occurs first, as assessed according to RECIST version 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (9):
- United States (5):
  - University of Colorado Denver Anschultz Medical Campus, Aurora, Colorado
  - Florida Cancer Specialists, Sarasota, Florida
  - Community Health Network, Indianapolis, Indiana
  - Start Midwest, Grand Rapids, Michigan
  - Swedish Cancer Institute, Seattle, Washington
- Spain (4):
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp Univ Fund Jimenez Diaz, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp Univ Hm Sanchinarro, Madrid

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency